CLINICAL TRIAL: NCT00279344
Title: A Randomised, Open, Parallel-group, Multi-centre Trial to Investigate Analgesic Efficacy and Safety of Transdermal Fentanyl (FITpatch) Compared to Standard Opioid Treatment in Cancer Pain.
Brief Title: Efficacy and Safety of FITpatch Compared to Standard Opioid Treatment in Cancer Pain (FT-015-IN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT-015-IN
Record Dates: First submitted 2005-12-14; First posted 2006-01-19 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Standard Opioid Analgesic Treatment of Cancer-related Chronic Pain.
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fentanyl (Matrifen)

SUMMARY:
Primary objectives:

* To determine non-inferiority of FITpatch with regard to efficacy compared to standard opioid treatment
* To assess the safety of FITpatch compared to standard opioid treatment

Secondary objectives:

* To assess the intake of oral morphine as rescue analgesic to FITpatch compared to standard opioid treatment
* To assess Quality of life reported with FITpatch compared to standard opioid treatment

ELIGIBILITY:
Inclusion Criteria:

Subjects that have insufficiently treated, cancer-related chronic pain that requires long-term treatment with an opioid at Step 3 on the WHO Ladder, and with Karnofsky performance status above 50.

1. Subject informed consent given.
2. Aged between 18 and 75 years, and for female subjects a proven negative pregnancy test and adequate contraception.
3. No significant skin lesions on relevant surfaces on the body or diffuse skin diseases.
4. No impaired respiratory function nor neurological or psychiatric impairment.
5. No known abuse of drug, narcotic or alcohol.
6. Not pregnant or nursing.
7. Not hypersensitive/allergic to fentanyl or morphine.
8. No head injury, primary brain tumor, increased intracranial pressure or impaired consciousness.
9. Not participating in other clinical trials.

Exclusion Criteria:

All exclusion criteria must be answered No for a patient to participate in the trial.

1. Does the patient have significant skin lesions on the upper arms/flat surface of the upper torso or diffuse skin disease (psoriasis or eczema) that preclude application of fentanyl patches?
2. Does the patient have a known abuse of drug, narcotic or alcohol?
3. Is the patient pregnant or nursing?
4. Has the patient neurological or mental impairment that may compromise data collection?
5. Is the patient hypersensitive/allergic to fentanyl or morphine or any of the ingredients in the trial medication?
6. Has the patient any major head injury, primary brain tumour, increased intracranial pressure or impaired consciousness?
7. Does the patient participate in other clinical with other investigational drugs or investigation al medical devices or has been participating in such a trial for the past 30 days?

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary:
To determine non-inferiority of FITpatch with regard to efficacy compared to standard opioid treatment and to assess the safety of FITpatch compared to standard opioid treatment

SECONDARY OUTCOMES:
Secondary:
To assess the intake of oral morphine as rescue analgesic to FITpatch compared to standard opioid treatment and to assess Quality of life reported with FITpatch compared to standard opioid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Project Management, Study Chair — Headquaters